CLINICAL TRIAL: NCT00765180
Title: Comparison of Transparent Retractable Extension Device and Narrow Band Imaging on Colorectal Adenoma Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TRE2
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal Cancer Screening
Keywords: colonoscopy; hood; NBI

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): The investigators evaluate beneficial effect of colonoscopy using narrow band imaging (NBI) for colorectal adenoma detection.
  Interventions: Device: TRE vs. NBI
- 1 (Experimental): The investigators evaluate the beneficial effect of colonoscopy with a transparent retractable extension (TRE) device on colorectal adenoma detection rate.
  Interventions: Device: TRE vs. NBI

INTERVENTIONS:
Device: TRE vs. NBI — TRE NBI

SUMMARY:
The investigators previously reported that colonoscopy with a transparent retractable extension (TRE) device improved the adenoma detection rate without affecting intubation and withdrawal times. On the other hand, colonoscopy using narrow band imaging (NBI) is expected to lead to higher rate s of adenoma detection. The investigators compared the effects of TRE device on colorectal adenoma detection with those of NBI.

ELIGIBILITY:
Exclusion Criteria:

* Age less than 20 years old
* Pregnant
* American Society of Anesthesiologists class III and IV
* Overweight (body weight > 100 kg)
* Allergic to the drugs used or its components (soybeans or eggs)
* Poor bowel preparation
* Previous colorectal surgical resection

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Colorectal adenoma detection rate | after colonoscopy

SECONDARY OUTCOMES:
Procedure time, complication | after colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan